CLINICAL TRIAL: NCT06791200
Title: Role of Some Biochemical Indices for Prediction of Acute Kidney Injury in Intensive Care Unit Patients in Upper Egypt
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ehdaa Ahmed Sanosy Mohamed, Ehdaa, Assiut University
Other Study IDs: prediction of AKI in icu
Record Dates: First submitted 2024-12-22; First posted 2025-01-24 (Actual); Last update posted 2025-01-24 (Actual); Status verified 2024-12

CONDITIONS: Acute Kidney Injury
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Diagnostic Test: biochemical indices — some biochemical indices for prediction of Acute kidney Injury

SUMMARY:
1. We will investigate the relation between the triglyceride-glucose index and the development of AKI in ICU.
2. To detect whether the TGI is a predictor of poor outcome (requirement of renal replacement therapy, or 14-day in-hospital mortality, and length of hospital stay) in ICU.
3. Compare TGL, Neutrophil-to-lymphocyte ratio, and clinical score (sequential organ failure assessment SOFA score) as predictors of poor outcome in ICU.

DETAILED DESCRIPTION:
Acute kidney injury (AKI) is a common clinical syndrome with a broad aetiological profile. It complicates about 5% of hospital admissions and 30% of admissions to intensive care units (ICU). During last 20 years has been a significant change in the spectrum of severe AKI such that it is no longer mostly a single organ phenomenon but rather a complex multisystem clinical problem. mortality from AKI, when part of MOF, remains over 50%.

In the past few decades, the understanding of AKI has greatly improved, but early diagnosis remains a great challenge. The performance of traditional kidney function index and serum creatinine is very limited for the early diagnosis of acute kidney injury The triglyceride glucose index (TGI) has been suggested as a useful marker of insulin resistance. Previous studies have shown that TGI is associated with many diseases, but no study has examined the relationship between TGI and Aki .

the primary objective of the present study was to investigate the relationship between TGI and Aki.

ELIGIBILITY:
Inclusion Criteria:

* The selected patients will be with the following inclusion criteria:

Patients admitted to ICU within 24 hours

Exclusion Criteria:

* We will exclude those with any of the following:

  1. Patients diagnosed more than 24 hours.
  2. Patients with missing data of triglyceride or glucose.
  3. Patients <18years old.
  4. patient with advanced liver disease and chronic kidney disease with or without dialysis

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The selected patients will be with the following inclusion criteria:
  Patients admitted to ICU within 24 hours
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-02-01 (Estimated); Primary Completion 2025-05-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
TGI | baseline

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Taghreed Sayed Mohamed Meshref s Meshref, Lecturer of Critical care med, Study Director — Assiut University
Locations (1):
- جامعة اسيوط, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Birkelo BC, Pannu N, Siew ED. Overview of Diagnostic Criteria and Epidemiology of Acute Kidney Injury and Acute Kidney Disease in the Critically Ill Patient. Clin J Am Soc Nephrol. 2022 May;17(5):717-735. doi: 10.2215/CJN.14181021. Epub 2022 Mar 15. PMID 35292532